CLINICAL TRIAL: NCT02748941
Title: Carotid Atherosclerosis : Innovative Imaging Biomarkers. Study Case-control
Acronym: ACABII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Fondation de France (Other); Bracco Imaging S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL15_0458
Record Dates: First submitted 2016-04-11; First posted 2016-04-22 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Carotid Stenosis
Keywords: unstable/stable atherosclerotic plaque; HITS; GSM; CEUS; HR MRI; mi-RNA
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- symptomatic and asymptomatic patients (Experimental)
  Interventions: Device: HITS quantification, Ultrasound examinations, High Resolution MRI

INTERVENTIONS:
Device: HITS quantification, Ultrasound examinations, High Resolution MRI — Simultaneously measure the occurrence of the event (ischemic stroke) and the characteristics of the atheromatous plaque
  Description of different modalities:
  HITS quantification
  Ultrasound examinations:
  * Ulceration >2 mm
  * Plaque thickness
  * GSM: computer analysis after normalization of most informative longitudinal view (image with maximum plaque area) using Photoshop
  * CEUS: plaque vascularization detection after bolus injection of SONOVUE on a video recording from the injection of the contrast (Vuebox - Bracco imaging)
  High Resolution MRI:
  * Stenosis severity, intraplaque hemorrhage, large lipid-rich necrotic core, ulceration or cap rupture and Brain MRI will be evaluated
  * Quantification of shear stresses (Pa) on the surface of the plaque
  mi-RNA identification and quantification

SUMMARY:
Cerebrovascular accident (CVA) constitutes a major health public problem. This represents the second cardiovascular death cause. CVA is ischemic in 80% of cases. Atheroma of large arteries, mainly carotid, is involved in about 20% of cases.

After several high grade studies (NASCET, ECST, ACAS, ACST), carotid surgery is based on stenosis calculation by Doppler ultrasound, CT angiography, MRI angiography or arteriography.

The composition of the plaque, showing its vulnerability, is associated with embolic risk and stroke. The therapeutic strategy based only on the narrowing of the arterial lumen is not satisfactory enough to prevent the occurrence of a transient ischemic attack (TIA) or an ipsilateral stroke due to carotid stenosis. Thus, new techniques emerge, to evaluate in vivo the inflammation of the plaque, its embolic consequences or the mechanical stress it undergoes. These techniques are: High Resolution MRI (HR MRI), evaluation of the Gray Scale Median (GSM) level, study of the plaque vascularization with Contrast Enhanced ultrasound (CEUS), High Intensity Transient Signals (HITS) by transcranial Doppler, micro RNA profile (mi RNA). These different modalities must be combined in order to increase the efficiency.

Based on these encouraging results, the investigator aim at evaluating the ability of different methods or their combination to predict the occurrence of ischemic stroke or TIA due to emboli from a carotid atherosclerotic plaque. Before considering a cohort study, he investigator want to evaluate the performance of each of these new methods in the characterization of carotid plaque instability. Performance evaluation will allow us to choose secondarily the most relevant association.

The investigator propose, as a first step, to make a case-control study with these methods, the cases are patients who had an ischemic stroke (authenticated by both the clinical exam and brain MRI) on the same side as the carotid stenosis and the controls are patients with carotid stenosis but without ischemic stroke. This study is a cross-sectional study because it simultaneously measures the occurrence of the event (ischemic stroke) and the characteristics of the atheromatous plaque.

Over a 2 year period, 45 symptomatic patients and 105 asymptomatic patients will be included with a carotid stenosis with at least a 50% caliber constriction according to NASCET criteria. (North American Symptomatic Carotid Endarterectomy Trial).

ELIGIBILITY:
Inclusion Criteria:

* Carotid stenosis ≥ 50% NASCET
* Case: ipsilateral carotid stenosis stroke, certified by MRI or CT in the preceding month, with no others causes of stroke
* Control: no clinical sign or MRI hint for a recent stroke
* Signed informed consent form
* Patient affiliated to a social security system or equivalent

Exclusion Criteria:

* Modified Rankin scale > 3
* Homolateral stroke or TIA > 1 month
* Medical history of homolateral carotid surgery, cervical radiation, carotid occlusive, homolateral intracranial stenosis, risk of developing arterial thromboembolic events
* Renal failure (creatinine clearance < 50 ml/min)
* Contraindication to ultrasound (sonovue)
* Contraindication to MRI and its contrast media (Gadolinium)
* Inability to sign informed consent
* Inability to undergo any of the technics (claustrophobia…)
* Serious co-morbid disease, dementia
* Neurological disease with no carotid disease
* Risk of pregnancy or pregnancy or breastfeeding
* Adult under reinforced guardianship or legal guardian
* Patient not understanding French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Number of HITS per hour in doppler ultrasonography | Day 1
Ulceration > 2 mm presence in doppler ultrasonography | Day 1
GSM (Gray Scale Median) quantification in doppler ultrasonography | Day 1
CEUS (Contrast Enhanced UltraSound ) | Day 1
  signal intensity amplification quantification and Ulceration > 2 mm
hemorrhage intra-plaque présence in HR MRI | Day 1
large lipid-rich necrotic core présence in HR MRI | Day 1
ulceration or cap rupture présence in HR MRI | Day 1

SECONDARY OUTCOMES:
hemorrhage intra-plaque | Day 1
  Compare the results of each modality for pathological analysis of the surgical equipment.
large lipid-rich necrotic core | Day 1
  Compare the results of each modality for pathological analysis of the surgical equipment.
ulceration or cap rupture | Day 1
  Compare the results of each modality for pathological analysis of the surgical equipment.
shear stresses (Pa) on the surface of the plaque | Day 1
  Quantification of the shear stresses (Pa) on the surface of the plaque with an analysis of hemodynamic environment using fluid dynamics mathematical models based on data collected by MRI.
mi-RNA identification | Day 1
  Identification of circulating mi-RNA specific to unstable atherosclerotic plaque by RT-PCR and comparison between case and control

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Service de radiologie, Bron, France

IPD SHARING:
Plan to Share IPD: No